CLINICAL TRIAL: NCT01466907
Title: Secondary Prevention and Health Promotion After Stroke A Nurse-led Randomized Controlled Open Trial
Brief Title: Secondary Prevention and Health Promotion After Stroke
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Skane University Hospital (Other)
Responsible Party: Principal Investigator, Ann-Cathrin Jonsson, Ass. Professor, Skane University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: MaStrokeFup0809; UMASNL (Other: Regional Ethical Review Board DNr 520/2007)
Record Dates: First submitted 2011-11-04; First posted 2011-11-08 (Estimated); Last update posted 2014-01-23 (Estimated); Status verified 2014-01

CONDITIONS: Stroke
Keywords: complication; depression; follow-up; intervention; nurse-led; outcome; secondary prevention; stroke
MeSH Terms: conditions — Stroke; Depression | interventions — Secondary Prevention

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention group (Active Comparator): Control of secondary prevention at three months and one year after stroke and referral to physician if medical interventions are needed. Assessment of functional status and self-reports on health outcome. Supportive counselling provided.
  Interventions: Other: Secondary prevention, supportive counselling
- Control group (Other): Standard care with no outlined follow-up until one year after stroke. Control of secondary prevention after one year after stroke and referral to physician if medical interventions are needed. Follow-up one year after stroke according to the same protocol as the intervention group.
  Interventions: Other: Standard care until one year follow-up

INTERVENTIONS:
Other: Secondary prevention, supportive counselling — Patients' self-reports on Mobility, Self Care, Usual activities, Pain/Discomfort, Anxiety/Depression, Health Outcome were registered. Health problems were assessed. Secondary prevention was controlled by measuring blood pressure, Cholesterol levels, HbA1c, Weight to estimate nutritional status. Functional status was assessed. Supportive counselling was provided. Referral was sent to physician if medical interventions were needed.
  Arms: Intervention group
Other: Standard care until one year follow-up — No intervention three months after stroke. Assessment one year after stroke and comparison with the intervention group.
  Arms: Control group

SUMMARY:
The aim of this study was to examine to what extent a one year population of stroke patients at a university hospital had well regulated risk factors and health problems one year after stroke, and if a structured nurse-led previous follow-up in the intervention group including referrals if needed could influence health outcome and risk factors one year after stroke.

DETAILED DESCRIPTION:
The follow-up protocol was categorized into Risk factors, Patients' self-reports, and Other health problems. Referral was sent to a physician if medical interventions were needed regarding risk factors measured above the limits as stated in the follow-up protocol in accordance with guidelines,and/or if any self-reported health problems were stated by the patients, or had been detected by the Specialist Nurse. Primary outcome was comparison between the intervention group and control group at one year after stroke regarding proportion of regulated risk factors, and self-reports on health outcome. Results of the two follow-ups of the intervention group were also compared.

ELIGIBILITY:
Inclusion Criteria:

WHO criteria for definition of stroke Signed consent

Exclusion Criteria:

Other diagnosis causing neurological symptoms

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 597 (Actual)
Dates: Start 2008-02; Primary Completion 2010-02 (Actual); Study Completion 2010-04 (Actual)

PRIMARY OUTCOMES:
Risk factors and health outcome compared between intervention group and control group | Baseline to one year after stroke for both groups.
  Outcome for both groups after one year was measured as the proportion of risk factors sufficiently treated, the patients' self-reports on health outcome and comparison between the intervention group and the control group.

SECONDARY OUTCOMES:
Risk factors and health outcome at two follow-ups. | Baseline to one year after stroke
  Comparison of health outcome at three months and one year after stroke in the intervention group.

CONTACTS AND LOCATIONS:
Overall Officials: Ann-Cathrin Jönsson, PhD, Principal Investigator — Department of Health Sciences, Lund University
Locations (1):
- Skåne University Hospital, Malmo, Sweden